CLINICAL TRIAL: NCT06368206
Title: Recording of Physiological Data Via an Optical Sensor At the Fingertip Alongside with Double Auscultatory and Pulse Oximetry to Evaluate the Effectiveness of an Optical Blood Pressure Monitoring (OBPM) Algorithm That Requires No Calibration with an External Cuff: a Single-center Prospective Clinical Study
Brief Title: Recording of Physiological Data Via an Optical Sensor At the Fingertip Alongside with Double Auscultatory and Pulse Oximetry to Evaluate the Effectiveness of an Optical Blood Pressure Monitoring (OBPM)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aktiia SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OBPM_Calfree2024
Record Dates: First submitted 2024-04-04; First posted 2024-04-16 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Blood Pressure

STUDY DESIGN:
Intervention Model Description: 1 study cohort that will test investigational device (Aktiia G2C) and Blood Pressure and Pulse Rate references.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Aktiia G2C and references/ comparators for Blood Pressure and Pulse Rate monitoring (Other): All study participants will test the investigational device (Aktiia G2C) and other marketed devices for blood pressure and pulse rate measurements (Aktiia Bracelet G2, Double auscultation, oscillometric monitors, finger pulse oximeter).
  Interventions: Device: Investigational device Aktiia G2C; Device: Marketed device used as reference for blood pressure monitoring: double auscultation cuff; Device: Marketed device used as comparative device for blood pressure and pulse rate monitoring: Aktiia Bracelet G2; Device: Marketed device used as comparative device for blood pressure and pulse rate monitoring: oscillometric upper-arm cuff; Device: Marketed device used as comparative device for blood pressure and pulse rate monitoring: oscillometric wrist cuff; Device: Marketed device used as reference for pulse rate monitoring: pulse finger oximeter

INTERVENTIONS:
Device: Investigational device Aktiia G2C — Study subjects are asked to stay seated and relaxed while successive measurements are taken with Aktiia G2C.
Device: Marketed device used as reference for blood pressure monitoring: double auscultation cuff — Study subjects are asked to stay seated and relaxed while successive measurements are taken with cuff for double auscultation.
Device: Marketed device used as comparative device for blood pressure and pulse rate monitoring: Aktiia Bracelet G2 — Study subjects are asked to stay seated and relaxed while successive measurements are taken with Aktiia Bracelet G2.
Device: Marketed device used as comparative device for blood pressure and pulse rate monitoring: oscillometric upper-arm cuff — Study subjects are asked to stay seated and relaxed while taking successive measurements with an oscillometric upper-arm cuff.
Device: Marketed device used as comparative device for blood pressure and pulse rate monitoring: oscillometric wrist cuff — Study subjects are asked to stay seated and relaxed while taking successive measurements with an oscillometric wrist cuff.
Device: Marketed device used as reference for pulse rate monitoring: pulse finger oximeter — Study subjects are asked to stay seated and relaxed while successive measurements are taken with pulse finger oximeter.

SUMMARY:
The present study, OBPM_Calfree2024, with N = 85 participants minimum over 1 visit (lasting around 1h), has been designed to collect raw optical data with Aktiia.product-G2C Clinical investigational system together with several reference systems within a cohort of subjects characterized by a wide variety of phenotypes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 21 to 85yo
* Subjects fluent in written and spoken French
* Subjects agreeing to attend the study visit and follow study procedures
* Subjects that have signed the informed consent form.

Exclusion Criteria:

* Amputated index fingers
* Damaged/injured skin at index fingers
* Damaged/injured skin at wrists
* Subjects suffering from sustained cardiac arrhythmias that can lead to weak or unstable pressure pulses including tachycardia (heart rate at rest > 120bpm) and atrial fibrillation
* Subjects suffering from pathologies that systematically reduce peripheral perfusion including Raynaud's disease, diabetes, renal dysfunctions (eGFR < 30mL/min/1.73 m2), hyper-/hypothyroidism, pheochromocytoma or arteriovenous fistula
* Pregnant women
* Polyneuropathy

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of study subjects that contribute with analyzable raw data collected | 1 hour
  Min 85 study subjects contribute with analyzable raw data collected

SECONDARY OUTCOMES:
Blood pressure mean value of differences | 1 hour
  The mean value of the differences between Aktiia G2C and double auscultation blood pressure measurements.
Blood pressure standard deviation of differences | 1 hour
  The mean value of the differences between Aktiia G2C and double auscultation blood pressure measurements.
Pulse rate root-mean-square error | 1 hour
  The root-mean-square difference between the Aktiia G2C pulse rate determinations and the reference method.

CONTACTS AND LOCATIONS:
Locations (1):
- CHUV, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No